CLINICAL TRIAL: NCT06183255
Title: New "System Medicine" Approach for the Development of Primary Prevention Strategies for Comorbidities in Infertile Men
Brief Title: "System Medicine" Approach for Prevention Strategies for Comorbidities in Infertile Men
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Salonia, Professor, IRCCS San Raffaele
Other Study IDs: RF-201912368847
Record Dates: First submitted 2023-12-05; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Infertility; Male Infertility
Keywords: Infertility; Male Infertility; Comorbidity
MeSH Terms: conditions — Infertility; Infertility, Male | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infertile men: Men with a diagnosis of pure Male Factor Infertility, as for WHO criteria
  Interventions: Other: Observation and evaluation of clinical parameters in the two cohorts
- Fertile men: Fathers with at least one child, spontaneously conceived, with a time-to-pregnancy within 12 months, as for WHO criteria
  Interventions: Other: Observation and evaluation of clinical parameters in the two cohorts

INTERVENTIONS:
Other: Observation and evaluation of clinical parameters in the two cohorts — During medical history evaluation, all factors that could negatively affect male fertility, like prevalent comorbidities, previous testis surgery, and any disorder affecting testicular function will be investigated in fertile and infertile men. Moreover, family history will be deeply investigated, including fertility status and prevalence of malignant Non Communicables Diseases. A comprehensive physical examination will be performed on each infertile and fertile man.

SUMMARY:
By applying a "system medicine" approach, the project aims to identify new biomarkers and/or prognostic tools aimed at developing personalized strategies to prevent the onset of comorbidities in infertile men.

DETAILED DESCRIPTION:
By applying a "system medicine" approach, the project aims to identify new biomarkers and/or prognostic tools aimed at developing personalized strategies to prevent the onset of comorbidities in infertile men.

The findings will provide new insights into the relationship between male infertility and somatic health, and shed light on the role of the microbiome in modulating the activity of the immune system. A "signature" of lack of immunological tolerance and biomarkers could be useful to predict future oncologic and non-oncological comorbidities in infertile men. This will let the development of a more clinically reliable and cost-effective personalized primary/secondary prevention strategy in a population at high risk of clinically relevant diseases.

ELIGIBILITY:
Inclusion Criteria:

* Signature of the informed consent;
* Be adults aged > 18;
* Caucasian race;
* Documented diagnosis of primary male infertility with pure male factor;

Exclusion Criteria:

* Failure to obtain informed consent;
* Patients with a known history of haematological disease;
* Patients undergoing antibiotic treatments in the last 6 months

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Fertile and infertile men according to WHO criteria (2010)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Medical anamnesis | Baseline
  Data collection on Charlson Comorbidity Index (CCI), partner's age, partner's health status;
Objective examination | Baseline
  presence of varicocele; testicular size and number
Testosterone | Baseline
  data on testosterone (ng/dL)
Genetic profile | Baseline
  Data on karyotype and microdeletions of the Y chromosome
Semen volume | Baseline
  Semen volume (ml)
Body mass index | Baseline
  Dataon Body mass index
Follicle-stimulating hormone | Baseline
  Data on follicle-stimulating hormone (mIU/ml)
Luteinizing hormone | Baseline
  Data on luteinizing hormone (mIU/dl)
Anti-Müllerian hormone | Baseline
  Data on Anti-Müllerian hormone (ng/ml)
Inhibin B | Baseline
  Data on Inhibin B (UI/mL)
Prolactin | Baseline
  Data on Prolactin (µg/l)
Thyroid-stimulating hormone | Baseline
  Data on thyroid-stimulating hormone (mU/L)
Osteocalcin levels | Baseline
  Data on osteocalcin levels (ng/ml)
Semen concentration | Baseline
  number of spermatozoa (million/ml)
Spermatozoa motility and morphology | Baseline
  motility and morphology of spermatozoa (%)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Salonia, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No